CLINICAL TRIAL: NCT00374621
Title: Randomized Clinical Trial of Cervical Ripening and Labor Induction Using Stepwise Oral Misoprostol With or Without Intravaginal Isosorbide Mononitrate
Brief Title: Trial of Cervical Ripening and Labor Induction Using Misoprostol With or Without Intravaginal Isosorbide Mononitrate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Yasser Yehia El-Sayed, Professor, Stanford University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 97274
Record Dates: First submitted 2006-09-07; First posted 2006-09-11 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Cervical Ripening
MeSH Terms: interventions — Misoprostol; isosorbide-5-mononitrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Misoprostol (Active Comparator)
  Interventions: Drug: Misoprostol with or without isosorbide mononitrate
- Misoprostol with Isosorbide Mononitrate (Active Comparator)
  Interventions: Drug: Misoprostol with or without isosorbide mononitrate

INTERVENTIONS:
Drug: Misoprostol with or without isosorbide mononitrate — Misoprostol 50 micrograms orally then 100 micrograms every 4 hours for up to four doses until modified Bishop score of 8 or higher was observed vs. the same misoprostol dosing plus isosorbide mononitrate 40 mg vaginally every 6 hours up to two doses total until a modified Bishop sore of at least 8 was observed

SUMMARY:
The purpose of this study is to determine the efficacy and safety of the addition of intravaginal isosorbide mononitrate to an established protocol of oral misoprostol for cervical ripening and labor induction.

ELIGIBILITY:
Inclusion Criteria::

* Pregnant women
* 18 years of age or greater
* Singleton pregnancy between 32-42 weeks gestation requiring labor induction
* Membranes must be intact

Exclusion Criteria:

* Ruptured membranes
* Gestational age less than 32 weeks
* Non-reassuring fetal heart rate tracing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2006-09; Primary Completion 2007-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Time to vaginal delivery | First dose of study medication to delivery

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Yehia El-Sayed, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Collingham JP, Fuh KC, Caughey AB, Pullen KM, Lyell DJ, El-Sayed YY. Oral misoprostol and vaginal isosorbide mononitrate for labor induction: a randomized controlled trial. Obstet Gynecol. 2010 Jul;116(1):121-126. doi: 10.1097/AOG.0b013e3181e408f2. PMID 20567177